CLINICAL TRIAL: NCT07010471
Title: A Phase 3, Randomized, Multi-Center, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Relutrigine in Participants With DEE Followed by an Open-Label Extension
Brief Title: A Clinical Trial for Participants With DEE to Assess Efficacy, Safety, Tolerability, and PK of Relutrigine
Acronym: EMERALD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRAX-562-311
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Developmental and Epileptic Encephalopathy 1
Keywords: DEE; Developmental and Epileptic Encephalopathy; epilepsy
MeSH Terms: conditions — Infantile Epileptic-Dyskinetic Encephalopathy; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Double-Blind Treatment Period (Experimental): Eligible participants will be randomly assigned in a double-blind manner and a 1:1 ratio to receive 1.0mg-1.5mg/kg relutrigine or placebo once daily orally or gastronomy/jejunostomy for 16 weeks
  Interventions: Drug: 1.0mg/kg/day PRAX-562; Drug: 1.5mg/kg/day PRAX-562
- Part A: Double-Blind Treatment Period (Placebo) (Placebo Comparator): Eligible participants will be randomly assigned in a double-blind manner and a 1:1 ratio to receive 1.0mg-1.5mg/kg relutrigine or placebo once daily orally or gastronomy/jejunostomy for 16 weeks
  Interventions: Drug: Placebo
- Part B: Open-Label Extension Treatment Period (Experimental): Participants from Part A will have the option to rollover to Part B to receive 1.0mg-1.5mg/kg of relutrigine once daily orally or gastronomy/jejunostomy for 32 weeks
  Interventions: Drug: 1.0mg/kg/day PRAX-562; Drug: 1.5mg/kg/day PRAX-562

INTERVENTIONS:
Drug: 1.0mg/kg/day PRAX-562 — Once daily orally or gastronomy/jejunostomy
  Other Names: relutrigine
  Arms: Part A: Double-Blind Treatment Period; Part B: Open-Label Extension Treatment Period
Drug: 1.5mg/kg/day PRAX-562 — Once daily orally or gastronomy/jejunostomy
  Arms: Part A: Double-Blind Treatment Period; Part B: Open-Label Extension Treatment Period
Drug: Placebo — Once daily orally or gastronomy/jejunostomy
  Arms: Part A: Double-Blind Treatment Period (Placebo)

SUMMARY:
A Phase 3, Randomized, Multi-Center, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Relutrigine in Participants with Developmental and Epileptic Encephalopathies Followed by an Open-Label Extension

ELIGIBILITY:
Inclusion Criteria:

* Has a documented diagnosis of a developmental and epileptic encephalopathy.
* Onset of seizures <12 years old.
* Has a weight >7 kg at the time of signing consent/assent.

Exclusion Criteria:

* Has a history of left bundle branch block, arrhythmias, Brugada syndrome, congenital heart disease, familial short QT syndrome, or family history of sudden death or ventricular arrhythmias, including idiopathic ventricular fibrillation.
* Had 2 or more episodes of convulsive status epilepticus requiring hospitalization and intubation in the 6 months prior to Screening.
* Has an abnormal ECG reading, including a QT interval corrected for heart rate using Bazett's method (QTcB) <350 and >450 ms (males), or <360 and >460 ms (females) at Screening and/or on Day 1.
* Any nerve stimulation must have been placed at least 3 months prior to Screening with at least 1 month of stable settings prior to Screening.
* Has received any other experimental or investigational drug, device, or other therapy within 30 days or 5 half-lives (whichever is longer) prior to Screening, including any prior use of gene therapy.
* Is currently pregnant or breastfeeding or is planning to become pregnant during the clinical trial or within 5 half-lives of the last study drug dose.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of relutrigine on seizure frequency in participants with DEEs compared to placebo | 16 weeks
  Change from baseline in monthly motor seizure frequency

SECONDARY OUTCOMES:
Achieve >50% reduction in monthly seizure frequency from baseline | 16 weeks
  Proportion of patients achieving >50% reduction in monthly seizure frequency from baseline
Change in seizure-free days | 16 weeks
  Change in seizure-free days from baseline
Clinical Global Impression-Severity questionnaire | 16 weeks
  CGI-S at baseline after 16 weeks
Clinical Global Impression-Improvement questionnaire | 16 weeks
  CGI-I subdomains scores after 16 weeks
Caregiver Global Impression-Severity questionnaire | 16 weeks
  CgGI-S at baseline after 16 weeks
Caregiver Global Impression-Improvement questionnaire | 16 weeks
  CgGI-I subdomains scores after 16 weeks
To evaluate the safety and tolerability of relutrigine in participants with DEEs | 16 weeks
  Incidence and severity of TEAEs
Columbia-Suicide Severity Rating Scale questionnaire | 16 weeks
  Incidence of suicidal ideation or behavior as measured by the C-SSRS
Evaluate the safety and tolerability of relutrigine in participants with DEEs | 16 weeks
  Incidence of clinically significant ECG abnormalities
To evaluate the safety labs and tolerability of relutrigine in participants with DEEs | 16 weeks
  The principal investigator (PI) or sub investigator will review the laboratory report and document this review. Any clinically significant adverse changes occurring during the clinical trial will be documented as adverse events.
To evaluate the change in respiratory rate and tolerability of relutrigine in participants with DEEs | 16 weeks
  Change in respiratory rate in breaths per minute
To evaluate the change in blood pressure and tolerability of relutrigine in participants with DEEs | 16 weeks
  Change in blood pressure in mm/Hg
To evaluate the change in pulse and tolerability of relutrigine in participants with DEEs | 16 weeks
  Change in heart rate in beats per minute
To evaluate the change in body temperature and tolerability of relutrigine in participants with DEEs | 16 weeks
  Change in tympanic temperature in Celsius

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Praxis Precision Medicines
Locations (5):
- United States (4):
  - Praxis Research Site, La Jolla, California
  - Praxis Research Site, Gulf Breeze, Florida
  - Praxis Research Site, Chevy Chase, Maryland
  - Praxis Research Site, Roseville, Minnesota
- Praxis Research Site, São Paulo, Brazil